CLINICAL TRIAL: NCT03883074
Title: Effect of a Combination Oral Formulation of Hyaluronic Acid With Chondroitin Sulphate and With Magnesium Trisilicate on Mucosal Integrity and Reflux Exposure in Subjects With Gastro-Esophageal Reflux Disease Not Currently Treated With a Proton Pump Inhibitor: a Double-Blind, Placebo-Controlled, Randomized, Crossover Study
Brief Title: Effect of a Combination of Hyaluronic Acid, Chondroitin Sulphate and Magnesium Trisilicate on Subjects With GastroEsophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PSC-DS TRIGERD 18
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GERDOff® Plus (Experimental): hyaluronic acid with chondroitin + sulphate + magnesium trisilicate Melt in mouth tablets (1100 mg). 1 tablet q.i.d. (three after meals, one before resting) for 3 consecutive weeks. After three weeks of wash-out period,patients will take either placebo or GERDOff® Plus q.i.d. (three after meals, one before resting) for another three weeks.
  Interventions: Device: hyaluronic acid with chondroitin + sulphate + magnesium trisilicate
- Placebo (Placebo Comparator): Placebo melt in mouth tablets (1100 mg). 1 tablet q.i.d. (three after meals, one before resting) for three consecutive weeks. After three weeks of wash-out period,patients will take either placebo or GERDOff® Plus q.i.d. (three after meals, one before resting) for another three weeks.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: hyaluronic acid with chondroitin + sulphate + magnesium trisilicate — Melt in mouth tablets (1100 mg)
  Other Names: GERDOff Plus
  Arms: GERDOff® Plus
Device: Placebo — tablets with the same aspect of the active device
  Other Names: Placebo (for hyaluronic acid with chondroitin + sulphate + magnesium trisilicate)
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate whether a 3-week treatment with an oral melt in mouth medical device, made up with hyaluronic acid, chondroitin sulphate and magnesium trisilicate, can lead to a reduction of Gastroesophageal Reflux Disease symptoms and to an improvement of the integrity of esophageal mucosa in patients who are to experiencing esophagus symptoms. The study is a randomized, double-blind cross-over placebo controlled study. Every patient will get both the active study device during one study period and placebo during another another period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 to 75 years
* GERD as defined by an acid exposure time >4% on pH/impedance monitoring and/or esophagitis LA grade A or B on endoscopy
* Heartburn at least twice per week over the last 1 month
* ReQuest Symptoms sum score >3,37 at screening
* GERD patients not treated with a PPI in the previous 2 months
* Subjects capable of understanding and be willing to provide signed and dated written voluntary informed consent

Exclusion Criteria:

* Patients suffering from gastrointestinal diseases other than GERD

  * Esophagitis LA grade C or D or Barrett's esophagus on endoscopy
  * Impaired kidney or liver function
  * Significant cardiac, pulmonary or psychiatric comorbidity as judged by the investigator
  * Medication use (including NSAIDS) that may interfere with GERD symptom assessment within 2 weeks before the start of the study or during the study
  * Pregnancy or breast-feeding
  * Females of childbearing potential in the absence of effective contraceptive methods
  * History of/or current psychiatric illness that would interfere with ability to comply with protocol requirements or give informed consent
  * History of alcohol or drug abuse that would interfere with ability to comply with protocol requirements
  * Treatment with any investigational drug within the previous 30 days
  * Active malignancy of any type, or history of cancer, including solid tumors and hematological malignancies (except patients with malignancies that have been surgically removed and/or with no evidence of recurrence for at least five years before study enrolment)
  * Inability to conform to protocol procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Esophageal Impedance | 3 weeks
  Change between groups in baseline impedance value. Impedance baseline values will be assessed in two steady periods of 30 seconds at the beginning and at the end of consecutive time windows of 30 minutes, 60 minutes.

SECONDARY OUTCOMES:
Esophageal acid exposure | 3 weeks
  Esophageal acid exposure assessed by 24-hour pH-impedance measurement
Esophageal permeability | 3 weeks
  Esophageal permeability assessed by transepithelial electrical resistance
Microscopic esophagitis | 3 weeks
  Microscopic esophagitis evidence at endoscopy assessed by Esohisto score. The score assesses the severity of esophagitis through a score for each parameter ranging from 0 to 2 (0=normal, 2=severe). Parameters are: Basal cell layer hyperplasia; Papillary elongation; Dilated intercellular spaces; Intraepithelial eosinophils; Intraepithelial neutrophils; Intraepithelial mononuclear cells
Intercellular spaces | 3 weeks
  The presence (on endoscopy) and severity of dilated intercellular spaces assessed by transmission electron microscopy.
The expression of tight junctions | 3 weeks
  The expression of tight junction proteins at RNA, protein and immunohistochemistry level
ReQuest Questionnaire score | 3 weeks
  Change in ReQuest score for GERD symptoms severity evaluated through ReQuest Questionnaire. ReQuest is a self-assessed, dimension-orientated scale designed to evaluate the treatment response in patients suffering from erosive GERD. It assesses seven dimensions of GERD (acid complaints, upper abdominal/stomach complaints, lower abdominal/ digestive complaints, nausea, sleep disturbances, other complaints and general well-being). The intensity is measured on a 100-mm visual analogue scale and the frequency (except general well-being) on a 7-point Likert scale, ranging from 0 to more than 10 times per day. It asks for the occurrence of symptom descriptions known to be typical of the corresponding dimension
Esophageal reflux episodes | 3 weeks
  Total number of reflux episodes and their proximal extent, number of acid reflux events and their duration.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Prof., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No